CLINICAL TRIAL: NCT06957067
Title: Reducing Dropout and Improving Outcomes From PTSD Therapy: When to Switch Therapies or Stay the Course
Acronym: STEER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: United States Department of Defense (U.S. Federal Agency)
Collaborators: University of Minnesota (Other); Lowcountry Center for Veterans Research (Unknown); Baylor College of Medicine (Other); Louisiana Veterans Research and Education Corporation (Unknown); Mayo Clinic (Other); Veterans Education and Research Association of Michigan (Unknown); Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency); Center for Veterans Research and Education (Other); New Orleans VA Medical Center (Unknown); Boston VA Research Institute, Inc. (Other); Arizona Veterans Research and Education Foundation (Unknown); Ocean State Research Institute, Inc. (Other); Veterans Education and Research Association of Northern New England, Inc (Unknown); Michael E. DeBakey VA Medical Center (U.S. Federal Agency); Phoenix VA Health Care System (U.S. Federal Agency); Charleston VA Medical Center (Unknown)
Responsible Party: Principal Investigator, Laura A. Meis, Principal Investigator, University of Minnesota
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 1806524-49; HT94252410639 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2025-03-28; First posted 2025-05-04 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-04

CONDITIONS: Post Traumatic Stress Disorder
Keywords: Cognitive Processing Therapy; Post Traumatic Stress Disorder; Trauma-focused treatments; Veterans
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Investigators will use a two-stage sequential, multiple assignment, randomized trial design (SMART) in which all participants beginning CPT are randomized to a first-stage intervention. In this first-stage, providers use one of two approaches to decision rules to identify patients who may be experiencing challenges in CPT (Catchall vs Targeted). The tailoring variables used in these decision rules will include weekly self-report measures and behavioral indicators. Investigators will evaluate if a participant meets criteria for their assigned decision rules every week during treatment. If individuals meet their decision rule criteria, participants will be randomized again to a second-stage intervention. For the second stage, providers will meet with their patients to either collaboratively consider switching to Present Centered Therapy or to discuss any problems they may be having with treatment using existing CPT skills, per randomization.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Catchall (Active Comparator): The Catchall approach to identifying individuals in need of intervention is intended to provide a generous, all-inclusive approach to identifying anyone who might have some concerns about their experiences with Cognitive Processing Therapy (CPT) and may benefit from discussing these concerns. The goal of this approach is to err on the side of intervening within anyone who may be experiencing challenges with the therapy. This approach assumes that spending a session talking about any concerns or struggles patients are having will help with patient-provider communication, improve attitudes about treatment, and improve treatment retention and outcomes.
  Interventions: Behavioral: Cognitive Processing Therapy; Behavioral: Measurement Based Care
- Targeted (Active Comparator): The Targeted approach to identifying individuals is intended to capture a narrower band of participants with clearer concerns about Cognitive Processing Therapy (e.g., at least one of their self-report scale scores is similar to or worse than patients who ultimately dropped out of CPT treatment in investigators' pilot data). Providers are more likely to miss some participants who may benefit from intervention through this approach but are less likely to unintentionally undermine CPT for participants who did not need intervention.
  Interventions: Behavioral: Cognitive Processing Therapy; Behavioral: Measurement Based Care
- CPT Skills (Active Comparator): Cognitive Processing Therapy is a 12-session, cognitive-behavioral treatment for PTSD that focuses on challenging and modifying maladaptive beliefs related to prior trauma. The goal is to build a new understanding of prior trauma in order to limit the negative influence trauma and it's reminders have on individuals' daily lives. CPT has built in strategies to address any challenges patients participating in the therapy. The degree to which these strategies are more effective than other approaches to addressing treatment challenges (e.g., switching to another therapy) are unknown.
  Interventions: Behavioral: CPT Skills; Behavioral: Cognitive Processing Therapy
- Consider Switching (Active Comparator): When patients are experiencing challenges with PTSD therapy, providers and their patients will consider switching from CPT to Present Centered Therapy. While PCT is somewhat less effective than CPT, it has solid evidence that it improves symptoms of PTSD. There is also no reflection on past trauma, homework demands are modest, and it has superior completion rates to CPT. Starting with a CPT and then considering switching to PCT, is a promising pathway to ensure individuals struggling in CPT complete an effective treatment. Given the efficacy differences between CPT and PCT, switching will be done collaboratively between patients and providers using shared decision making (versus requiring all patients to switch to PCT). This ensures the choice to switch is patient-centered and relevant to how these decisions would be made in real-world care.
  Interventions: Behavioral: Cognitive Processing Therapy; Behavioral: Present Centered Therapy; Behavioral: Shared Decision Making

INTERVENTIONS:
Behavioral: CPT Skills — CPT trainings recommend that if an individual is experiencing challenges with the CPT protocol (e.g., ambivalence about continuing treatment or struggling with completing homework), the provider can apply the skills of CPT to that particular problem. Those skills include problem solving and cognitive restructuring to identify and alter maladaptive underlying beliefs. The purpose of this work is to address the individual's underlying problem or problematic beliefs to improve the individual's attitudes about CPT and/or improve the individual's compliance with treatment activities. The therapist's end-goal is to keep the individual moving forward in the CPT protocol.
  Arms: CPT Skills
Behavioral: Cognitive Processing Therapy — CPT is a 12-session, cognitive-behavioral treatment for PTSD that focuses on challenging and modifying maladaptive beliefs related to prior trauma. The goal is to build a new understanding of prior trauma in order to limit the negative influence trauma and it's reminders have on individuals' daily lives. The treatment involves education about PTSD and skill building to identify and challenge maladaptive, trauma-related thinking through Socratic questioning and worksheets that teach individuals to challenge this thinking themselves. Later sessions focus on specific themes that are difficult for individuals with PTSD and can keep individuals "stuck" in their symptoms. Themes include safety, trust, control, self-esteem, and intimacy.
  Although the skills utilized in CPT may be used to respond to challenges individuals have with participating in CPT, the effectiveness of these strategies has not been explicitly tested.
Behavioral: Present Centered Therapy — PCT was developed as a comparator for "active" TFT, so protocol length typically matches the comparator. PCT focuses on "current life problems as manifestations of PTSD" in weekly 60-minute sessions. It includes psychoeducation and normalization of responses to trauma, problem solving related to life difficulties and stress, and emotional support and validation. Its hypothesized mechanisms are increased interpersonal connection and mastery in managing life stressors. Therapist skills include validation, support, and reflective listening. The first 2 sessions provide an overview and rationale for PCT. Subsequent sessions focus on topics participants choose and are less structured. Participants use a daily diary to record any concerning problems or issues they experience during the week. These diaries are used to select session topics.
  Arms: Consider Switching
Behavioral: Shared Decision Making — Shared decision making (SDM) is widely considered the best model for achieving patient-provider agreement on treatment plans and an ethical imperative for decision making. SDM is a communicative process in which patients and their provider personalize treatment approaches to the individual, their situation, and the problems that they are experiencing. Providers and patients engage in a shared deliberation of meaningful treatment alternatives, including pros and cons, how choices align or misalign with values, and patients' abilities to complete the plans under consideration.
  Arms: Consider Switching
Behavioral: Measurement Based Care — Investigators will compare methods of identifying individuals experiencing challenges in CPT. Investigators will use self-report measures administered each week during treatment to identify individuals who may be struggling in during CPT and compare two approaches to cut scores on these measures to classify individuals as "in need of intervention." Investigators will also use behavioral indices to determine if veterans are in need of intervention, including homework compliance and session attendance. One approach will liberally classify many individuals as "in need of intervention" (Catchall), while the other will take a more targeted approach (Targeted).
  Arms: Catchall; Targeted

SUMMARY:
Investigators' overall objective is to compare methods of identifying individuals who may be experiencing challenges in Cognitive Processing Therapy (CPT) and compare methods of intervening to optimize treatment retention and outcomes. Investigators' specific aims are:

1. to determine whether the use of CPT skills versus collaboratively considering switching to Present Centered Therapy (PCT) is more effective in improving outcomes for individuals experiencing challenges with CPT. Outcomes include post-traumatic stress disorder (PTSD) severity [primary], depression, functioning, and treatment retention;
2. to compare two approaches to identifying individuals in CPT in need of additional support during treatment;
3. to study the barriers and facilitators of implementing these intervention strategies.

Finally, exploratory aims will examine the stability of differences between treatment conditions, compare combinations of interventions tested, and examine moderators of intervention effects.

DETAILED DESCRIPTION:
Background: Trauma-focused treatments (TFTs) for PTSD, including Cognitive Processing Therapy (CPT), result in clinically significant symptom relief for many. However, they are not equally effective for everyone, and an important subgroup will discontinue before fully completing therapy. Identifying this subgroup is an important, but elusive, first step. In their prior work, investigators found Veterans were often unlikely to tell providers about the nature and extent of the challenges they experienced while trying to effectively participate in TFTs. Use of behavioral and attitudinal indices that do not rely on individuals' willingness to speak up in session may help providers identify with whom to intervene. Using weekly measures, investigators will compare two approaches to cut scores to classify individuals as "in need of intervention." One will liberally classify many individuals (Catchall); the other will take a more targeted approach (Targeted). For the present study, investigators will focus on CPT, as it is the most widely disseminated TFT in VA and DoD.

Once investigators have used the above approaches to identify individuals who may need additional support and help with CPT, an important next question is what is the most effective way to intervene with these individuals. TFTs have built in strategies for flexing the treatments to help patients who are experiencing challenges in treatment. These strategies are of unknown efficacy. Alternatively, patients and their therapists could consider switching to a different form of therapy besides TFTs. Present Centered Therapy (PCT) may be a well-suited alternative. While PCT is somewhat less effective than TFTs, it has solid evidence of efficacy. There is no reflection on past trauma, homework demands are modest, and it has superior completion rates to TFTs. Starting with CPT and then considering switching to PCT, is a potentially promising pathway to ensure individuals who are challenged by CPT complete an effective treatment. Given the efficacy differences between CPT and PCT, switching should be done collaboratively between patients and providers (versus forcing all participants to PCT). This ensures the choice to switch is patient-centered, relevant to real-world care, and consistent with Veteran end-users' recommendations.

Objectives/Aims: Investigators overall objective is to compare methods of identifying individuals who may be experiencing difficulties with CPT and compare methods of intervening to optimize treatment retention and outcomes. Investigators will use weekly measures developed with Veteran end-users to identify individuals who could benefit from intervention. When identified, providers will either use CPT skills to address participants' treatment challenges or collaboratively consider switching to PCT.

Investigators' specific aims are:

1. to determine whether the use of CPT skills versus collaboratively considering switching to PCT is more effective in improving outcomes for individuals experiencing challenges with CPT. Outcomes include PTSD severity [primary], depression, functioning, and treatment retention;
2. to compare two approaches (Catchall versus Targeted) to identifying individuals in CPT in need of additional support;
3. to study the barriers/facilitators of implementing these intervention strategies.

Finally, exploratory aims will examine the stability of differences, compare combinations of interventions tested, and examine moderators of intervention effects.

Study Design: Investigators propose a sequential multiple assignment randomized trial (SMART) where investigators first randomize 280 CPT patients to one of the two approaches to identify who needs extra support in CPT (Catchall vs Targeted). Participants deemed "in need of intervention" will then be randomized again to either (a) CPT skills or (b) to collaboratively consider switching. Outcomes will be assessed using structured clinical interviews (PTSD severity) and self-report (functioning and depression) at baseline, posttreatment, 3-, and 6-months posttreatment. Investigators will also study the implementation of their interventions through a mixed methods process evaluation. The study treatment with Veteran participants will take place across four VAs (Houston, Charleston, New Orleans, and Phoenix) over 4-years.

Clinical Impact: Investigators expect to learn an optimal approach to identifying individuals who need extra support during CPT and an optimal approach for addressing their needs. This will help ensure all individuals reach their maximal potential in PTSD treatment. The proposed work addresses multiple sub-areas within FY23 TBIPHRP CTA Focus Area 3 (Treat) through adapting or combining interventions so they can achieve their greatest impact on the lives and functioning on Service Members and Veterans, promoting sustained functional recovery, and enhancing the relevance of research to practice via hybrid effectiveness implementation studies.

Relevance to Military Health: The influence of a successful course of PTSD treatment on an individual's life is considerable. In addition to reducing PTSD and associated mental health symptoms (e.g., depression), successful PTSD treatment reduces suicidal ideation and improves, reduces, and may even reverse the negative physical health effects associated with the disorder. Yet, abundant heterogeneity remains in therapy response. Investigators propose using rigorous methods to alter CPT mid-stream to ensure that PTSD treatment promotes recovery from PTSD for more Service Members. Investigators will also explore differences for women, an important priority for the DoD. This work is essential for moving the science of therapy forward. To investigators' knowledge, this will be the first to study to test a strategy for considering switching from trauma to non-trauma focused therapies. Such research is critical to military service retention and to the health of the entire military. Findings from this work will yield an evidence base for personalizing PTSD treatment to make it more tolerable and more effective for more people.

ELIGIBILITY:
Inclusion Criteria:

* Veterans interested in outpatient VA psychotherapy for PTSD
* Meets DSM-5 criteria for PTSD
* Be able to provide informed consent
* Be willing to be randomized
* Agree to not receive non-study psychotherapy for PTSD during study treatment (case management, supportive therapy/group, and concurrent substance use treatment are allowable)

Exclusion Criteria:

* Severe cognitive impairment
* Current suicidal or homicidal intent with a specific plan
* Uncontrolled psychotic or manic symptoms
* A psychiatric medication change in the past month
* A severe SUD as diagnosed by the DSM-5

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
PTSD severity (via structured clinical interview) | Baseline, through six-months after treatment completion. Treatment completion takes an average of 4 months.
  Measured using the Clinician-Administered PTSD Scale for the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (CAPS-5). This standardized interview is conducted by an evaluator blinded to study condition, via telehealth.

SECONDARY OUTCOMES:
Depression severity | Baseline, through six-months after treatment completion. Treatment completion takes an average of 4 months.
  Self-report surveys using established, validated instruments will be used to assess secondary outcomes. In routine care, CPT response is typically evaluated through repeated PHQ-9 administration, rather than through structured clinical interview. Thus, these self-reports will be administered to facilitate comparisons with outcomes in real-world care. They will also be used by clinicians for monitoring treatment response and determining treatment end-date.
PTSD severity (via self report) | Baseline, through six-months after treatment completion. Treatment completion takes an average of 4 months.
  Self-report surveys using established, validated instruments will be used to assess secondary outcomes. In routine care, CPT response is typically evaluated through repeated PCL-5 administration, rather than through structured clinical interview. Thus, these self-reports will be administered to facilitate comparisons with outcomes in real-world care. They will also be used by clinicians for monitoring treatment response and determining treatment end-date.
Psychosocial functioning (IPF scores) | Baseline, through six-months after treatment completion. Treatment completion takes an average of 4 months.
  Self-report surveys using established, validated instruments will be used to assess secondary outcomes. For psychosocial functioning, investigators will assess individuals' self-reported functioning on the Inventory of Psychosocial Functioning (IPF). The IPF is a self-report instrument developed specifically for assessing PTSD-related functional impairment. The instrument measures each of the PTSD-related functional domains determined to matter most to individuals with PTSD: relationships with intimate partners, family relationships, work performance, friend relationships, parenting, educational performance, and self-care functioning (e.g., maintaining personal hygiene, exercising, household chores, healthy eating). The total scale will be used, which is the average of the total number of subscales of relevance to the respondent (i.e., respondent skips employment functioning items if they are not employed).
Treatment completion | At the end of treatment. Treatment takes an average of 4 months.
  Participants will be considered to have completed treatment if they complete the final session of their treatment protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Meis, PhD, Principal Investigator — Women's Health Sciences Division of the National Center for PTSD; University of Minnesota; Princess Ackland, PhD, Principal Investigator — University of Minnesota
Locations (4):
- United States (4):
  - VA Phoenix Health Care System, Phoenix, Arizona
  - New Orleans VA Medical Center, New Orleans, Louisiana
  - Ralph H. Johnson VA Health Care System (Charleston VA), Charleston, South Carolina
  - VA Houston Healthcare System, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Study data will be reported only in aggregate in any reports or publications; no names of study participants will be used in any reports or publications resulting from this study. In accordance with 38 USC 7332, this type of information will be kept confidential and will not be disclosed in presentations, publications, or any other dissemination of the study results, or to anyone outside of the IRB-approved study team. Deidentified datasets will be made available following study completion. Participants will be notified of this during informed consent.
Supporting Information: Study Protocol

REFERENCES:
- [Background] Bradley R, Greene J, Russ E, Dutra L, Westen D. A multidimensional meta-analysis of psychotherapy for PTSD. Am J Psychiatry. 2005 Feb;162(2):214-27. doi: 10.1176/appi.ajp.162.2.214. PMID 15677582
- [Background] Steenkamp MM, Litz BT, Hoge CW, Marmar CR. Psychotherapy for Military-Related PTSD: A Review of Randomized Clinical Trials. JAMA. 2015 Aug 4;314(5):489-500. doi: 10.1001/jama.2015.8370. PMID 26241600
- [Background] Maguen S, Li Y, Madden E, Seal KH, Neylan TC, Patterson OV, DuVall SL, Lujan C, Shiner B. Factors associated with completing evidence-based psychotherapy for PTSD among veterans in a national healthcare system. Psychiatry Res. 2019 Apr;274:112-128. doi: 10.1016/j.psychres.2019.02.027. Epub 2019 Feb 11. PMID 30784780
- [Background] Nahum-Shani I, Almirall D, Yap JRT, McKay JR, Lynch KG, Freiheit EA, Dziak JJ. SMART longitudinal analysis: A tutorial for using repeated outcome measures from SMART studies to compare adaptive interventions. Psychol Methods. 2020 Feb;25(1):1-29. doi: 10.1037/met0000219. Epub 2019 Jul 18. PMID 31318231
- [Background] Meis LA, Polusny MA, Kehle-Forbes SM, Erbes CR, O'Dougherty M, Erickson EPG, Orazem RJ, Burmeister LB, Spoont MR. Making sense of poor adherence in PTSD treatment from the perspectives of veterans and their therapists. Psychol Trauma. 2023 May;15(4):715-725. doi: 10.1037/tra0001199. Epub 2022 Mar 24. PMID 35324228
- [Background] Lei H, Nahum-Shani I, Lynch K, Oslin D, Murphy SA. A "SMART" design for building individualized treatment sequences. Annu Rev Clin Psychol. 2012;8:21-48. doi: 10.1146/annurev-clinpsy-032511-143152. Epub 2011 Dec 12. PMID 22224838
- [Background] Maguen S, Holder N, Madden E, Li Y, Seal KH, Neylan TC, Lujan C, Patterson OV, DuVall SL, Shiner B. Evidence-based psychotherapy trends among posttraumatic stress disorder patients in a national healthcare system, 2001-2014. Depress Anxiety. 2020 Apr;37(4):356-364. doi: 10.1002/da.22983. Epub 2019 Dec 18. PMID 31850650
- [Background] Kehle-Forbes SM, Ackland PE, Spoont MR, Meis LA, Orazem RJ, Lyon A, Valenstein-Mah HR, Schnurr PP, Zickmund SL, Foa EB, Chard KM, Alpert E, Polusny MA. Divergent experiences of U.S. veterans who did and did not complete trauma-focused therapies for PTSD: A national qualitative study of treatment dropout. Behav Res Ther. 2022 Jul;154:104123. doi: 10.1016/j.brat.2022.104123. Epub 2022 May 21. PMID 35644083
- [Background] Meis LA, Noorbaloochi S, Hagel Campbell EM, Erbes CR, Polusny MA, Velasquez TL, Bangerter A, Cutting A, Eftekhari A, Rosen CS, Tuerk PW, Burmeister LB, Spoont MR. Sticking it out in trauma-focused treatment for PTSD: It takes a village. J Consult Clin Psychol. 2019 Mar;87(3):246-256. doi: 10.1037/ccp0000386. PMID 30777776
- [Background] Howard KP, Spoont MR, Polusny MA, Eftekhari A, Rosen CS, Meis LA. The role of symptom accommodation in trauma-focused treatment engagement and response. J Trauma Stress. 2023 Jun;36(3):524-536. doi: 10.1002/jts.22912. Epub 2023 Feb 13. PMID 36782380
- [Background] Belsher BE, Beech E, Evatt D, Smolenski DJ, Shea MT, Otto JL, Rosen CS, Schnurr PP. Present-centered therapy (PCT) for post-traumatic stress disorder (PTSD) in adults. Cochrane Database Syst Rev. 2019 Nov 18;2019(11):CD012898. doi: 10.1002/14651858.CD012898.pub2. PMID 31742672
- [Background] Holliday R, Holder N, Monteith LL, Suris A. Decreases in Suicide Cognitions After Cognitive Processing Therapy Among Veterans With Posttraumatic Stress Disorder Due to Military Sexual Trauma: A Preliminary Examination. J Nerv Ment Dis. 2018 Jul;206(7):575-578. doi: 10.1097/NMD.0000000000000840. PMID 29905663